CLINICAL TRIAL: NCT03914846
Title: Clinical Implementation of a Novel Ultrasound Technology for the Evaluation of Skin Lesions and Sentinel Lymph Node
Brief Title: Ultrasound in Diagnosing Patients With Skin Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Mohammad K. Khan, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB00086913; NCI-2019-01754 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RAD4512-18 (Other: Emory University Hospital/Winship Cancer Institute)
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Skin Lesion
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort I (ultrasound) (Experimental): Patients with skin lesions undergo at least 1 ultrasound during the consultation. Patients may undergo at most 2 additional scans after the standard of care approach for non-malignant lesions at the discretion of the radiation oncologist and/or dermatologist.
  Interventions: Procedure: Ultrasound
- Cohort II (ultrasound) (Experimental): Skin cancer patients who undergo surgery or radiation undergo 2-5 ultrasounds over a 1 year period (a baseline ultrasound scan may be performed prior to treatment, followed by 1 scan during and/or after radiation, and additional ultrasounds may be conducted [at the discretion of the treating physician] upon completion of radiation and/or surgery, at approximately 1, 6, and 12 month follow-up examinations).
  Interventions: Procedure: Ultrasound
- Cohort III (ultrasound) (Experimental): Participants with inflammatory skin disorders (psoriasis, eczema, alopecia, acne) undergo ultrasound at baseline and follow-up visits.
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Undergo ultrasound with elastography

SUMMARY:
This trial studies the use of a novel non-invasive ultrasound technique in diagnosing patents with skin lesions. Diagnostic procedures, such as ultrasound, may be a less invasive way to check skin lesions for skin cancer and other skin disorders.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Characterize a wide variety of lesions including but limited to:

I a. Malignant lesions: basal cell cancers, squamous cell cancers, Merkel cell cancer, melanoma, etc.

I b. Non-malignant lesions: keloids, surgical scars, actinic keratosis, benign and dysplastic nevi, cysts, lipoma.

I c. Inflammatory conditions: psoriasis, eczema, alopecia, acne, wounds, etc). I d. Determine if ultrasound can be used to more effectively/accurately administer treatment (injections, surgical procedures, etc).

II. Characterize pre and post treatment changes in the lesion as well as the surrounding normal tissue stroma (examples, but not limited to: changes to hair follicles, epidermis, dermis, subcutaneous tissue, erector pillae muscles, vessels, nerves, etc).

III. Correlate ultrasonographic findings with histological findings for lesions that would have been removed surgically and/or are biopsied (examples, but not limited to: removal of a skin cancer where ultrasound is used to characterize peripheral extent of the lesion as well as depth of penetration, a benign versus malignant lesion, pigmented versus [vs] non-pigmented lesion, etc).

IV. Determine if ultrasound can be used to monitor acute and late toxicity. V. See if ultrasound can also image sentinel lymph nodes that may potentially contain cancer.

OUTLINE: Patients are assigned to 1 of 3 cohorts.

COHORT I: Patients with skin lesions undergo at least 1 ultrasound during the consultation. Patients may undergo at most 2 additional scans after the standard of care approach for non-malignant lesions at the discretion of the radiation oncologist and/or dermatologist.

COHORT II: Skin cancer patients who undergo surgery or radiation undergo 2-5 ultrasounds over a 1 year period (a baseline ultrasound scan may be performed prior to treatment, followed by 1 scan during and/or after radiation, and additional ultrasounds may be conducted [at the discretion of the treating physician] upon completion of radiation and/or surgery, at approximately 1, 6, and 12 month follow-up examinations).

COHORT III: Participants with inflammatory skin disorders (psoriasis, eczema, alopecia, acne) undergo ultrasound at baseline and follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Candidate with skin lesions.
* Signed study-specific informed consent prior to study entry.

Exclusion Criteria:

* Prior surgery or radiotherapy to the area to be treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Pre and post treatment changes in lesions | 12 months from study start
  Ultrasound findings will be reviewed for changes in lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad K. Khan, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No